CLINICAL TRIAL: NCT00923468
Title: ADVL08N1: A Pharmacokinetic Participation Questionnaire Study
Brief Title: Pharmacokinetic Studies Participation Survey
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080223; 08-C-0223
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-31

CONDITIONS: Relapsed Solid Tumors; Relapsed Leukemia; Relapsed Brain Tumors
Keywords: Pharmacokinetics; Phase I Trials; Children; Relaspsed Solid Tumors; Relapsed Leukemia; Relapsed Brain Tumors
MeSH Terms: conditions — Leukemia; Brain Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* A pharmacokinetic (PK) study of a new drug involves taking several blood samples over a period of time from study participants to determine how the body handles the substance. These studies provide critical information about new drugs.
* Often, patients or parents of children in drug studies choose not to participate in optional PK studies that are part of the study protocol.
* A better understanding of why patients or families do or do not agree to participate in PK studies may help researchers make it easier for people to participate in them.

Objectives:

* To learn why some people do or do not agree to participate in PK blood sampling studies.

Eligibility:

* Patients 18 years of age and older and parents or guardians of children who are participating in a study of a drug that includes the option of participating in PK sampling.

Design:

* Participants fill out a 2-page survey asking about why they did or did not participate in the study's PK sampling.

DETAILED DESCRIPTION:
Background:

Pharmacokinetic studies provide critical information about the disposition of anticancer drugs in children. However, participation of children in the pharmacokinetic portion of phase I studies is optional when there is not prospect of direct benefit to the child.

The rate of participation in optional PK studies on COG Phase I Consortium Studies has been 60-70%.

There are no recent data on why families do or do not agree to participate in optional PK studies. Understanding families' reasons may reveal barriers to participation that could be overcome, leading to increased participation rates in optional PK sampling.

Objectives:

To use a simple 2 page survey to gather preliminary information on why parents/children agree to participate in Phase I Studies do or do not agree to participate in the voluntary pharmacokinetic (PK) portion of those studies.

Eligibility:

Subjects (greater than or equal to 18 years old) or parents/guardians of subjects who are minors who consented to Phase I studies with optional PK sampling with the previous 4 weeks.

Consent for the primary Phase I treatment protocol must be active (not withdrawn).

No limit on the number of prior Phase I studies in which the subject or subject's child participated.

Subjects may only participate in this study once.

Design:

The individual who provided consent to the treatment study that included optional PK sampling will complete a short questionnaire.

Subjects (n=50) from a convenience sample will complete and return the questionnaire.

Reasons for participating or agreeing to participate will be tabulated. Correlations between answers and subject demographics, time required by PK, need for additional IV will be sought.

Subjects will meet off study criteria when the questionnaire is returned, lost to follow up, or consent for data submission to this or the primary treatment protocol is withdrawn.

The total accrual is 50 subjects. Accrual ceiling at the POB, NCI is 25 subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects who consented within the 4 weeks prior to enrollment on this questionnaire study to a Phase 1 study that included optional PK sampling. (If the subject was a minor and a parent or legally authorized representative provided consent, subject for this questionnaire study refers to the parent). The PK questionnaire should be completed within 4 weeks of when the subject consented to the study that included optional PK sampling. (Note: The Phase 1 study need not have been a COG study).
* Subjects are eligible regardless of whether they initially agreed to participate in the PK portion and regardless of whether they actually completed the PK sampling (as long as reason for not completing the sampling was not withdrawal of consent).
* Subjects must not have withdrawn consent to the study that included optional PK sampling.
* Subjects must not have initially agreed to optional PK sampling but then withdrawn consent for sampling prior to completing the questionnaire.
* Subjects are eligible regardless of how many phase 1 or other studies they have enrolled in the past.
* Each subject may participate only once in the survey.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2008-09-23; Primary Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States